CLINICAL TRIAL: NCT03881163
Title: Phase I Study to Evaluate Pharmacokinetics, Safety and Tolerability of Single and Multiple i.v. Doses of N-acetylcysteine (NAC) in Chinese Healthy Volunteers
Brief Title: A Study to Evaluate Pharmacokinetics, Safety and Tolerability of Single and Multiple Intravenous Doses of N-acetylcysteine (NAC) in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Z7244J01
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Tract Disorders
MeSH Terms: conditions — Respiration Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: All the subjects enrolled in the study will receive the same treatment with the investigational medicinal product (IMP), i.e. NAC, 300 mg/ 3 mL solution injection as single dose and multiple dose regime. Single dose of IMP will be administered under fasting conditions on day 1 at 08:00 ±1 h. Multiple doses (5) of IMP will be administered twice a day (b.i.d.) on days 4 and 5 at 08:00 ±1 h and 20:00 ±1 h and one dose will be administered on day 6 at 08:00 ±1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose regime of N-acetylcysteine (NAC) (Experimental): On day 1 at 08:00 ±1 hours, one dose of 600 mg of NAC (300 + 300 mg ampoule) will be administered under fasting conditions.
  Interventions: Drug: N-acetylcysteine (NAC)
- Multiple dose regime of N-acetylcysteine (NAC) (Experimental): On days 4 and 5 at 08:00 ±1 hours and 20:00 ±1 hours and at 08:00 ±1 on day 6, 5 doses of 600 mg of NAC (300 + 300 mg ampoule) will be administered.
  Interventions: Drug: N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — Two ampoules of IMP (300 + 300 mg) corresponding to a total dose of 600 mg of NAC diluted in 10 mL of NaCl 0.9% sterile saline solution, will be administered by a 5-minute i.v. infusion.

SUMMARY:
This is a single and multiple dose, single centre, open-label, one-way, pharmacokinetics, safety and tolerability clinical trial of Phase I to be performed in Chinese healthy male and female volunteers. Twenty-four (24) healthy male and female Chinese volunteers will be included in the study. Drop-out subjects will not be replaced. The study has been designed in agreement with the Chinese Technical Guideline on Clinical Pharmacokinetic Research of Chemical Drugs, 18 March 2005 and the European Guideline on the Investigation of Bioequivalence. No randomisation will take place in this study. All the participant will receive the same treatment with the investigational medicinal product (IMP), i.e. NAC, 300 mg/ 3 mL solution for injection.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Ethnicity, Sex and Age: Chinese males and females, 18-45 year old inclusive
3. Weight: body weight ≥50 kg
4. Body Mass Index: 19-26 kg/m2 inclusive
5. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting/supine position
6. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
7. Nicotine addiction (smoker subjects only): ability to abstain from smoking for the duration of the clinical study
8. Contraception and fertility (women only): women of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 60 calendar days before the screening visit
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 60 calendar days before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner

Women of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. Women of childbearing potential should be willing to adopt abstinence or contraception measures during the study and two weeks post-dose. For all women, pregnancy test result must be negative at screening and day -1.

Exclusion Criteria:

1. Electrocardiogram (12-lead ECG in supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness, in particular significant laboratory abnormality indicative of hepatic condition (more than 3 times the upper limit)
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, urologic, metabolic, neurological or psychiatric diseases, as determined by the investigator, that may interfere with the aim of the study; history of carcinoma in situ and malignant disease; active bacterial or viral infection and fever >38°C within 48 h prior to study treatment administration
6. Virology: positive result of HIV, hepatitis B (HBV), hepatitis C (HCV) or Treponema pallidum (TP) assays
7. Surgery: any surgery within 60 calendar days of screening (excluding diagnostic surgery)
8. Medications: medications, including over the counter (OTC) medications, herbal remedies and traditional Chinese remedies for 2 weeks before the start of the study. Hormonal contraceptives for women will be allowed
9. Investigative drug studies: participation in the evaluation of any investigational product for 1 month before this study
10. Blood donation: blood donations for 90 calendar days before this study
11. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015-2020] caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
12. Abuse drug test: positive urine abuse drug test at screening or day -1
13. Alcohol test: positive alcohol breath test at day -1
14. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians; consumption of alcohol, grapefruit, products containing grapefruit, or beverages containing xanthines (coffee, tea, soda, coffee with milk, energy drinks) within 48 hours prior to the enrolment
15. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women
16. Vaccination within 4 weeks of study treatment
17. Other unspecified reasons that, in the opinion of the investigator, make the subject unsuitable for enrolment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, No.197 Ruijin Er Road, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a single center study conducted in China from 11 November 2019 to 18 January 2020. All participants randomized in the study received single and multiple doses of N-acetylcysteine (NAC).
Pre-assignment Details: Participants who met the eligibility criteria at the Screening Visit (Day -14 to Day 1) were assigned to receive NAC.
Groups:
- Overall - NAC 600 mg: All participants were dosed with NAC once daily (QD) at 08:00 ± 1 hour on Day 1 under fasting conditions, twice daily (BID) at 08:00 ± 1 hour and 20:00 ± 1 hour on Day 4 and Day 5 after one 3-day wash-out, and QD at 08:00 ± 1 hour on Day 6.
Period: Overall Study
Arm/Group | Overall - NAC 600 mg
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Overall - NAC 600 mg: All participants were dosed with NAC QD at 08:00 ± 1 hour on Day 1 under fasting conditions, BID at 08:00 ± 1 hour and 20:00 ± 1 hour on Day 4 and Day 5 after one 3-day wash-out, and QD at 08:00 ± 1 hour on Day 6.
Arm/Group | Overall - NAC 600 mg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (5.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 24
Region of Enrollment [Number; unit: participants]
  China | 24

OUTCOME MEASURES:

1. Primary Outcome: Peak Drug Concentration (Cmax) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single administration of the investigational product.
Time Frame: On Day 1 and Day 2-At pre-dose (0) and 5 (at the end of the infusion), 8, 12, 15, 20, 25, 30, 60 minutes and 2, 4, 6, 8, 10, 12, 24 and 32 hours post-dose
Population: Pharmacokinetic (PK) set: all enrolled participants who fulfilled the study protocol requirements in terms of investigational medicinal product intake and had evaluable PK data readouts for the planned analyses, with no major deviations that might affect the PK results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Single Dose - NAC 600mg: Participants who met the eligibility criteria at the Screening Visit were assigned to receive NAC. On day 1 at 08:00 ±1 hours, one dose of 600 mg of NAC (300 + 300 mg ampoule) was administered under fasting conditions.
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
µg/mL | 83.30 (30.7)

2. Primary Outcome: Time to Achieve Cmax (Tmax) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
hours | 0.083 [0.08 to 0.25]

3. Primary Outcome: Terminal Elimination Rate Constant (Kel) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
1/hour | 0.09723 (56.8)

4. Primary Outcome: Half-life (t1/2) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
hour | 7.129 (56.8)

5. Primary Outcome: Area Under the Concentration-time Curve (AUC) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
h*µg/mL
  AUC from time zero to the last observed concentration time t [AUC(0-t)] | 87.16 (17.4)
  AUC extrapolated to infinity [AUC(0-inf)] | 93.94 (18.0)
  AUC from time zero to 12 hours post-dose [AUC(0-12h)] | 81.87 (14.0)

6. Primary Outcome: Volume of Distribution (Vd) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
litre | 65.69 (44.8)

7. Primary Outcome: Total Body Clearance (CLt) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter\hour
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
Liter\hour | 6.387 (18.0)

8. Primary Outcome: Total Amount of NAC Excreted in Urine [Ae(0-t)] After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
μg
  Ae(0-4) | 62750 (76.4)
  Ae(4-8) | 16170 (55.2)
  Ae(8-12) | 3609 (155.0)
  Ae(12-24) | 1846 (78.0)
  Ae(24-32) | 1366 (63.9)
  Ae(0-8) | 84020 (53.4)
  Ae(0-12) | 89600 (50.5)
  Ae(0-24) | 92020 (49.4)
  Ae(0-32) | 93490 (48.5)

9. Primary Outcome: Total Fraction of NAC Dose Excreted in Urine [Fe(0-t)] After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fraction
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
fraction
  Fe(0-4) | 0.1046 (76.4)
  Fe(0-8) | 0.1400 (53.4)
  Fe(0-12) | 0.1493 (50.5)
  Fe(0-24) | 0.1534 (49.4)
  Fe(0-32) | 0.1558 (48.5)

10. Primary Outcome: Renal Clearance (CLr) After Single Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
mL/h | 995.2 (50.2)

11. Primary Outcome: Percentage of the AUC(0-inf) Obtained by Extrapolation (%AUCextra)
Description: To evaluate pharmacokinetic parameters of NAC in plasma after single dose administration of the investigational product.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Single Dose - NAC 600mg
Number analyzed (Participants) | 24
percentage | 6.967 (26.8)

12. Primary Outcome: Plasma Concentration at Steady-state After Multiple Doses of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after multiple dose administration of the investigational product.
  Css_max = maximum NAC plasma concentration at steady-state, Css_min=minimum plasma concentration at steady-state, Css_avg=average NAC plasma concentration at steady-state.
Time Frame: On Day 4 and Day 5 -At pre-dose. On Day 6 and Day 7-At pre-dose (0) and 5 (at the end of the infusion), 8, 12, 15, 20, 25, 30, 60 minutes and 2, 4, 6, 8, 10, 12, 24 and 32 hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Multiple Dose - NAC 600mg: Participants who met the eligibility criteria at the Screening Visit were assigned to receive NAC. On days 4 and 5 at 08:00 ±1 hours and 20:00 ±1 hours and at 08:00 ±1 on day 6, 5 doses of 600 mg of NAC (300 + 300 mg ampoule) will be administered.
Arm/Group | Multiple Dose - NAC 600mg
Number analyzed (Participants) | 24
µg/mL
  Css_max | 100.8 (29.1)
  Css_min | 1.899 (20.9)
  Css_avg | 7.719 (14.1)

13. Primary Outcome: Time to Achieve Css_max (tss_max) After Multiple Doses of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after multiple dose administration of the investigational product.
Time Frame: as for outcome 12
Population: Pharmacokinetic (PK) set: all participants who fulfilled the study protocol requirements in terms of investigational medicinal product intake and had evaluable PK data readouts for the planned analyses, with no major deviations that might affect the PK results.
Measure: Median (Full Range); unit: hour
Arm/Group | Multiple Dose - NAC 600mg
Number analyzed (Participants) | 24
hour | 0.083 [0.07 to 0.13]

14. Primary Outcome: Area Under the Concentration-time Curve at Steady State After Multiple Doses of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after multiple dose administration of the investigational product.
  AUCss(0-12h)=AUC at steady-state from the last multiple dose to 12 hours post-dose, AUCss(0-t)=AUC at steady-state from the last multiple dose to the last observed concentration time t.
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Multiple Dose - NAC 600mg
Number analyzed (Participants) | 24
h*µg/mL
  AUCss(0-t) | 116.6 (15.1)
  AUCss(0-12h) | 92.63 (14.1)

15. Primary Outcome: Accumulation Ratio After Multiple Doses of NAC
Description: as for outcome 13
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Multiple Dose - NAC 600mg
Number analyzed (Participants) | 24
Ratio | 1.132 (6.0)

16. Primary Outcome: Total Amount of NAC Excreted in Urine From the Last Multiple Dose to 32 h at Steady-state [Aess(0-32)]
Description: as for outcome 13
Time Frame: as for outcome 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | Multiple Dose - NAC 600mg
Number analyzed (Participants) | 24
μg | 68980 (68.1)

17. Primary Outcome: Degree of Fluctuation Over One Dosing Interval at Steady-state (DF%) After Multiple Dose of NAC
Description: To evaluate pharmacokinetic parameters of NAC in plasma after multiple dose administration of the investigational product.
  Degree of fluctuation over one dosing interval at steady-state is calculated as (Css_max - Css_min)/ Css_av*100
Time Frame: as for outcome 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Multiple Dose - NAC 600mg
Number analyzed (Participants) | 24
percentage | 1279 (30.7)

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: To collect safety and tolerability data after single and multiple dose administration of the investigational product.
Time Frame: From screening to Final Visit/early termination visit (ETV, Day 8)
Population: Safety set: All participants who received at least one dose of investigational medicinal product.
Measure: Count of Participants; unit: Participants
Groups:
- NAC 600 mg: All participants were dosed with NAC once daily (QD) at 08:00 ± 1 hour on Day 1 under fasting conditions, BID at 08:00 ± 1 hour and 20:00 ± 1 hour on Day 4 and Day 5 after one 3-day wash-out, and QD at 08:00 ± 1 hour on Day 6.
Arm/Group | NAC 600 mg
Number analyzed (Participants) | 24
Participants
  Any TEAE | 7
  Any TEAE Related to investigational medicinal product | 2

ADVERSE EVENTS:
Time Frame: From Screening to Final Visit/Early termination (ETV, Day 8)
Description: All AEs/serious adverse events (SAEs), regardless of the relationship to investigational medicinal product, were to be assessed and recorded from the date the informed content form was signed until Final Visit/ETV.
Groups:
- Overall - NAC 600 mg: All participants were dosed with NAC once daily (QD) at 08:00 ± 1 hour on Day 1 under fasting conditions, BID at 08:00 ± 1 hour and 20:00 ± 1 hour on Day 4 and Day 5 after one 3-day wash-out, and QD at 08:00 ± 1 hour on Day 6.
Arm/Group | Overall - NAC 600 mg
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 7/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall - NAC 600 mg (N=24)
Urine output increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Weight decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03881163/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT03881163/SAP_001.pdf